CLINICAL TRIAL: NCT04206423
Title: Grip Strength or Pinch Strength: Which is Preferred to Evaluate Lateral Epicondylitis?
Brief Title: Grip Strength or Pinch Strength in Lateral Epicondylitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif GÜLER, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREH9
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Lateral Epicondylitis
Keywords: Disability evaluation; Hand Strength; Quality of life; Pain; Pinch Strength; Tennis elbow
MeSH Terms: conditions — Tennis Elbow; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Age and sex matched healthy controls
- Lateral epicondylitis: Newly diagnosed lateral epicondylitis patients.
  1. Pain in lateral epicondylitis region
  2. Pain increase with palpation
  3. Positivity in two diagnostic test out of three (Maudley's test, Mill's test or Cozen's test)

SUMMARY:
Grip strength can be decreased in lateral epicondylitis. Pinch strength is also affected in people suffering from lateral epicondylitis. In this study, participants will be evaluated using a hydraulic dynamometer, a pinch meter and we will evaluate pain, disability and quality of life.

DETAILED DESCRIPTION:
Newly diagnosed patients with lateral epicondylitis and healthy controls will be included in the study with an allocation ratio of 2:1. Using a hydraulic dynamometer grip strength will be evaluated three times, one minute between each measurement. Then palmar pinch, key pinch and tip pinch measurements will be evaluated for three times each. For each measurement, the participants will rest one minute between repetitive measurements, and five minutes between each parameters. The order of measurements will be randomized for each participants to avoid bias. Then the participants will be evaluated using different scales for pain, disability and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pain in elbow for at least two weeks

Exclusion Criteria:

* Nonsteroidal antiinflammatory drug usage during last week.
* Rheumatic diseases (Rheumatoid arthritis, systemic lupus erythematosus, reactive arthritis, etc.)
* Malignancy
* Extracorporeal shock wave therapy in last six months
* Lateral epicondylitis injection in last six months or any treatment.
* Lateral epicondylitis brace usage

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants suffering from lateral epicondylitis will be included in the patient group and healthy control will be included in control group.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Hand (grip) Strength | 0.day
  Maximum and Pain free hand grip strength using a handheld dynamometer
Pinch Strength (key pinch, palmar pinch and tip pinch) | 0.day
  Maximum and Pain free hand grip strength using a handheld dynamometer

SECONDARY OUTCOMES:
Visual Analog Scale (VAS)-During day | 0.day
  Pain during day will be evaluated using visual analog scale
VAS-Night | 0.day
  Pain during night will be evaluated using visual analog scale
Patient Rated Tennis Elbow Evaluation Scale | 0.day
  The questions will help to understand the amount of difficulty the patient have had with their arm in the past week. The patient will be describing their average arm symptoms over the past week on a scale 0-10.
Disability | 0.day
  The Disabilities of the Arm, Shoulder and Hand Scale
World Health Organization-Quality of Life- Bref (WHOQOL-BREF) scale | 0.day
  The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Y Yalcınkaya, Ass. Prof., Study Chair — Gaziosmanpasa Training and Research Hospital
Locations (1):
- Gaziosmanpasa Taksim Research and Education Hospital, Istanbul, Turkey (Türkiye)